CLINICAL TRIAL: NCT02588807
Title: The Combination of Phospholipids and Medical Herbs for the Treatment of Patients With Amyotrophic Lateral Sclerosis (ALS); A Pilot Study
Brief Title: Food Supplement for the Treatment of Patients With Amyotrophic Lateral Sclerosis
Acronym: ALS-PHL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor and hospital did not reach agreement
Sponsor: Herb Spirit (Industry)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0015-14-CMC
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spirit1 (Experimental): Patients will take a daily nutritional supplement for 8 months
  Interventions: Drug: Spirit1

INTERVENTIONS:
Drug: Spirit1 — Spirit 1 is a combination of phospholipids and anti-oxidant medicinal plants

SUMMARY:
The purpose of the study is to evaluate the safety of combining phospholipids with medicinal plants for treatment of patients with amyotrophic lateral sclerosis (ALS)

DETAILED DESCRIPTION:
This is an open label pilot study, where patients (n=10) with ALS will take a daily nutritional supplement for 8 months. After documenting the ALS symptom history at baseline, the disease severity, and the motor muscles functions will be assessed at baseline and every two months (0, 2 , 4, 6, 8 months of the treatment). Adverse events and side effect will be assessed on every visit and throughout the experiment. In addition, the level of renal function, liver function and electrolytes will be evaluated from blood samples taken at baseline, 4, and 8 months visits.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 to 75 years, Females>50 years
2. Diagnosis of "probable" or "definite" ALS according to the El Escorial revised criteria
3. A documented history of ALS symptoms for more than 6 month prior to study enrolment, and no more than 40 month.
4. Patients capable of understanding and signing Informed Consent.

Exclusion Criteria:

1. Patients allergic to seafood
2. Patients with forced vital capacity < 75%
3. Patients who are respiratory dependent, underwent tracheostomy, or cannot swallow.
4. Patients with cardiovascular diseases
5. Patients with diabetes
6. Patients with active peptic ulcers
7. Diagnosis of other neurodegenerative diseases (Parkinson disease, Alzheimer disease, etc).
8. Patients suffering from other chronic significant disease, malignant diseases or any other disease that may risk the patient or interfere with the ability to interpret the results.
9. Patients that can not sign/understand the Informed Consent Form.
10. Female patients who are pregnant or lactating
11. Patients who have received and experimental drug or have participated in a clinical trial within 1 month prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Tolerability and safety based on the number and severity of adverse events (AE) | 8 months
  Tolerability and safety evaluations will be based on the documentation of the incidence and severity of short term, and long term side effects, and adverse events (AEs) as well as changes in results of blood tests (increase in levels of liver enzymes, decrease in renal function, changes in complete blood count and electrolytes).

SECONDARY OUTCOMES:
Change from baseline in score on the ALS Functional Rating Scale Revised (ALS-FRSr) | 4, 8 months
  The ALS-FRS-R is an instrument for evaluating the activities of daily living and global function of patients with ALS. It is used to monitor functional change in a patient over time and includes 12 questions. Each question has 5 possible responses (0-indicates unable to 4-indicates normal ability). Individual item scores are added to produce a reported score of between 0 = worst and 48 = best.
  A change of ≥25% is considered a clinically meaningful deterioration.
Change from baseline in Forced vital capacity (FVC) | 2, 4, 6, 8 months
  The purpose of this test is to assess the extent of respiratory muscle fatigue. The amount and/or speed (volume and flow respectively) of air that can be inhaled and exhaled will be measured by a commercial spirometer. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation.
Change from baseline in hand grip power using a dynamometer | 2, 4, 6, 8 months
  The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles. The subject holds a commercial dynamometer in the hand to be tested, with the arm at right angles and the elbow by the side of the body. When ready the patient will be asked to squeezes the dynamometer with maximum force which is maintained for 3 seconds. This will be repeated 3 times in each hand. The best result from several trials for each hand is recorded, with at least 15 seconds recovery between each effort.
Change from baseline in walking speed for 10 meters | 2, 4, 6, 8 months
  The purpose of this test is to measure the lower extremities muscle strength. The patients will be asked to walk a distance of 10 meters in their maximal speed. The time to walk this distance will represent the lower extremities muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Meer, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Hacarmel Hospital, Haifa, Israel